CLINICAL TRIAL: NCT04026958
Title: Antibiotic-mediated Improvements in Vigilance: Mechanisms of Action of Clarithromycin in Hypersomnia Syndromes
Brief Title: Clarithromycin Mechanisms in Hypersomnia Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Lynn Marie Trotti, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00108681; 1R01NS111280 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Narcolepsy Without Cataplexy; Idiopathic Hypersomnia; Narcolepsy With Cataplexy
Keywords: Neurology
MeSH Terms: conditions — Idiopathic Hypersomnia; Narcolepsy | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clarithromycin (Experimental): Participants in this study arm will receive clarithromycin for 14 days.
  Interventions: Drug: Clarithromycin
- Placebo (Placebo Comparator): Participants in this study arm will receive a placebo to match clarithromycin for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clarithromycin — Clarithromycin will be dosed as 500 mg twice daily, once upon awakening and once with lunch, for 14 days.
  Other Names: Biaxin
  Arms: Clarithromycin
Drug: Placebo — A placebo to match clarithromycin will be dosed as 500 mg twice daily, once upon awakening and once with lunch, for 14 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate a medication called clarithromycin for treating sleepiness in narcolepsy and idiopathic hypersomnia. Studies have shown that clarithromycin can reduce sleepiness, but researchers do not know how clarithromycin does this. This study will look at brain activity (on magnetic resonance imaging [MRI]), inflammation, bacteria living in the gut, and cerebrospinal fluid, to better understand how clarithromycin can reduce sleepiness. This study will recruit 92 participants who will be randomized to receive clarithromycin or a placebo for 14 days.

DETAILED DESCRIPTION:
Excessive daytime sleepiness and long sleep durations are common features of many neurologic disorders, including myotonic dystrophy, Parkinson's disease, and the central nervous system hypersomnia syndromes.

Pathologic daytime sleepiness in the central nervous system hypersomnia disorders impairs occupational performance, limits quality of life, and more than doubles motor vehicle and other accident risk. Because the underlying cause of the majority of these hypersomnia syndromes is not known, treatments are aimed at increasing monoaminergic signaling involved in wake promotion. Yet, at least one-fourth of patients with hypersomnia syndromes cannot achieve satisfactory control of symptoms with these treatments and disability or medical leaves of absence are often necessary. There is a clear need for novel treatments for excessive daytime sleepiness to resolve this failure of the current standard of care.

In prior studies, clarithromycin resulted in significant, clinically meaningful improvements in sleepiness severity, sleepiness-related limitations in extended activities of daily living, and sleepiness-related quality of life. Long sleep durations and sleep inertia, both ancillary symptoms of hypersomnia disorders that contribute to functional impairments, were also improved with clarithromycin.

Hypothesis: Clarithromycin will reduce excessive sleepiness and other symptoms of hypersomnia disorders, as measured by self-report and objective testing.

Aim 1: To identify central nervous system mediators of clarithromycin's ability to promote wakefulness and reduce sleepiness, among patients with central hypersomnia syndromes.

Hypothesis 1a: Changes in cerebrospinal fluid (CSF) enhancement of gamma-aminobutyric acid-A (GABA-A) receptor function in vitro will be associated with improvements in self-reported and objectively measured sleepiness.

Hypothesis 1b: Changes in functional connectivity will be associated with improvements in self-reported and objectively measured sleepiness.

Aim 2: To probe extra-neuronal mechanisms by which clarithromycin may reduce sleepiness, including changes in systemic inflammation and changes in gastrointestinal microbiota composition, in patients with central hypersomnia syndromes.

Hypothesis 2a: Improvement in sleepiness with clarithromycin use will be positively associated with reductions in systemic inflammation, especially reductions in levels of tumor necrosis factor-alpha (TNFα).

Hypothesis 2b: Improvement in sleepiness with clarithromycin use will be positively correlated with modulation of gastrointestinal dysbiosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic hypersomnia or narcolepsy
* age 18-60
* free of wake-promoting medication, sleepy despite current wake-promoting medications, or willing to discontinue current wake-promoting medication for at least 5 half-lives prior to baseline measures

Exclusion Criteria:

* other potential causes of hypersomnolence, including untreated moderate or severe sleep apnea, severe periodic limb movement disorder with arousals, uncontrolled metabolic disorders
* contraindication to clarithromycin
* contraindication to any of the study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Epworth Sleepiness Scale Score | Day -1, Day 14
  The Epworth Sleepiness Scale asks participants to respond to 8 scenarios with how likely they are to fall asleep on a 4-point scale where 0 = "would never doze" and 3 = "high chance of dozing". Total scores range from 0 to 24 where higher scores indicate a higher chance of falling asleep during daytime activities.
Change in Maintenance of Wakefulness Test (MWT) | Day -1, Day 14
  The MWT polysomnographic procedure examines how well participants stay awake during several trials where participants relax in a quiet room for 40 minutes. One study found the mean sleep latency among persons without a sleep disorder to be 35.2 minutes. Sleep latency is compared between study arms.
Change in gamma-aminobutyric acid receptor A (GABA-A) potentiation | Day -1, Day 14
  Cerebrospinal fluid (CSF) is drawn to determine the change in levels of GABA-A potentiation between the study arms. The difference between measured current with GABA alone and the current measured with GABA + CSF yields a measure of potentiation for each CSF sample in each condition.
Change in Default Mode Network (DMN) Connectivity | Day -2, Day 13
  The default mode network (DMN) consists of a group of highly correlated brain regions most active during quiet rest. DMN connectivity changes with sleep states and it is increasingly implicated in the symptomatology of sleepiness. During resting state, sleep deprived participants demonstrate reduced static connectivity with the DMN. Changes in DMN between the Baseline 1 and Day 13 visits are compared between treatment groups, particularly using quasi-periodic patterns (QPPs), which interrogate network-level connectivity on a dynamic scale. Preservation of the temporal dimension provides more insight into how this spatiotemporal network propagates across condition and pathology.
Change in tumor necrosis factor - alpha (TNF-α) | Day -1, Day 14
  Blood samples are used to determine the change in levels of TNF-α between the study arms. TNF-α is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in gastrointestinal microbiome composition | Day -1, Day 14
  Changes in microbiome composition via 16S ribosomal ribonucleic acid (rRNA) sequencing results are compared between study arms.

SECONDARY OUTCOMES:
On-Treatment Sleep Duration | Day -1, Day 14
  Participants log when they go to bed and when they wake up in order to calculate the number of minutes spent sleeping. The average duration of sleep across 14 days is compared between study arms.
Change in Fatigue Severity Scale (FSS) Score | Day -1, Day 14
  Fatigue severity is measured with the Fatigue Severity Scale (FSS). The FSS is a 9-item instrument where responses are on a scale of 1 to 7 where 1 = "disagree" and 7 = "agree". Total scores range from 9 to 63 where higher scores indicate greater fatigue.
Change in Multidimensional Fatigue Inventory (MFI-20) Score | Day -1, Day 14
  The MFI-20 is a 20-item instrument assessing fatigue severity. Responses are on a 5-point scale where 1 = "yes, that is true" and 5 = "no, that is not true". Positively phrased items are reverse scored so that the total score ranges from 20 to100 where higher scores indicate greater severity of fatigue.
Change in Sleep Inertia Questionnaire (SIQ) Score | Day -1, Day 14
  The SIQ is an instrument with 21 items with responses on a 5-point scale where 1 = "not at all" and 5 = "all the time". Two additional questions relate to how much time it takes for the respondent to wake up in the morning. Total scores range from 21 to 105 and higher scores indicate increased difficulty from tiredness.
On-Treatment Sleep Inertia Likert Scale | Day -1, Day 14
  Sleep inertia is measured with a single item on a 10-point Likert scale asking participants how difficult it was for them to wake up in the morning, where 1 = "not difficult at all" and 10 = "very difficult". The average scores across 14 days are compared between study arms.
Change in Interleukin 1 alpha (IL-1α) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-1α between the study arms. IL-1α is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Interleukin 1 beta (IL-1β) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-1β between the study arms. IL-1β is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Interleukin 2 (IL-2) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-2 between the study arms. IL-2 is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Interleukin 6 (IL-6) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-6 between the study arms. IL-6 is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Interleukin (IL-8) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-8 between the study arms. IL-8 is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Interleukin (IL-15) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-15 between the study arms. IL-15 is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Interleukin (IL-18) | Day -1, Day 14
  Blood samples are used to determine the change in levels of IL-18 between the study arms. IL-18 is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in tumor necrosis factor beta (TNF-β) | Day -1, Day 14
  Blood samples are used to determine the change in levels of TNF-β between the study arms. TNF-β is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in interferon alpha (INF-α) | Day -1, Day 14
  Blood samples are used to determine the change in levels of INF-α between the study arms. INF-α is a soporific cytokine and a reduction in soporific cytokines is hypothesized to reduce daytime sleepiness.
Change in Functional Outcomes of Sleep Questionnaire (FOSQ) Score | Day -1, Day 14
  The FOSQ is a 30-item instrument assessing how sleepiness impacts daily activities. There are five subscales assessing General Productivity, Activity Level, Vigilance, Social Outcomes, and Intimate and Sexual Relationships. Items are scored on a 4-point scale where 1 = extreme difficulty and 4 = no difficulty. Subscale scores are obtained by calculating the mean score for the items in that subscale and each can range from 1 to 4, where higher scores indicate less difficulty due to sleepiness. A total score is obtained by calculating the means of the subscale scores and multiplying that by the number of subscales with a score. The total score ranges from 5 to 20 and higher scores indicate fewer difficulty from sleepiness.
Change in Hypersomnia Severity Index (HSI) | Day -1, Day 14
  The HSI is a 9-item instrument assessing the severity of excessive sleepiness (hypersomnolence). Items are scored on a Likert scale where 0 = not at all and 4 = very much. Total scores range from 0 to 36 and higher scores indicate greater severity of symptoms of hypersomnia.
Change in MRI Functional Connectivity | Day -2, Day 13
  For functional connectivity analyses, each functional scan is parceled into the 246 regions of interest (ROIs) contained in the Brainnetome Atlas and mean timecourse is calculated for each ROI. Pearson correlations between each pair of ROIs are calculated, to determine the strength of functional connectivity between each pair of regions. This yields a functional connectivity matrix for each functional scan (at both a subject- and group-level). These correlation matrices are Fischer z-transformed and averaged across each condition to create a mean functional connectivity matrix for each condition.
Change in MRI Activation Patterns | Day -2, Day 13
  Participants complete a working memory task during functional magnetic resonance imaging (fMRI). The change in task performance (accuracy and reaction time for 0-back, 1-back, and 2-back tasks) from baseline to on-treatment is compared between conditions. Activity during the task (vs non-task) is calculated for each participant within regions of interest defined by prior meta-analysis identifying areas involved in this working memory task. Activation in these areas at baseline will be compared to activation on study treatment, and differences between clarithromycin and placebo groups compared. QPPs will also be used to further probe these task-associated differences.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Marie Trotti, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Emory Sleep Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
After de-identification, individual patient data collected during the trial that underlie the results reported in the article will be available to be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 3 months after article publication and ending 3 years after article publication. Reasonable attempts will be made to accommodate requests after 3 years.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, and with other entities who provide a clear rationale for data use. Data will be shared for analyses to achieve the aims of the approved proposal. Proposals for using the data should be directed to lbecke2@emory.edu.

DOCUMENTS (1):
  • Informed Consent Form (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04026958/ICF_000.pdf